CLINICAL TRIAL: NCT05265377
Title: Safety and Usability of the STELO Exoskeleton in People With Acquired Brain Injury and Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Centro de Referencia Estatal de Atención Al Daño Cerebral (Other); National Research Council, Spain (Other Government); Centro Lescer (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STELO-US_DCA+LM
Record Dates: First submitted 2022-01-11; First posted 2022-03-03 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injury; Acquired Brain Injury
Keywords: exoskeleton; modular; SCI; ABI; gait; spinal cord injury; acquired brain injury
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STELO Exoskeleton (Experimental): 3 treatment sessions will be performed with the Stelo exoskeleton.
  Interventions: Device: Stelo

INTERVENTIONS:
Device: Stelo — Use of Stelo exoskeleton in nine rehabilitation sessions

SUMMARY:
Gait impairment in people with acquired brain injury (ABI) and spinal cord injury (SCI) can be very heterogeneous. For this reason, STELO has been developed: a new concept of exoskeleton based on modular technology for gait assistance. It allows a personalised configuration according to the functional capacity of each patient, as the therapist can choose which robotic joints to use depending on the therapeutic goal and on the patient recovery phase. The objective is to analyse the usability of the STELO modular exoskeleton in people with ABI and SCI.

DETAILED DESCRIPTION:
A test phase will be conducted in healthy volunteers as a proof of concept with the aim of evaluating safety and usability in healthy participants prior to the use of the device in the ABI or SCI population (Phase 2).

After verifying that the device is safe in healthy people, phase 2 will begin: it consists of a total of 10 visits. These visits will include gait training sessions using the STELO modular exoskeleton.

ELIGIBILITY:
Inclusion Criteria:

* Weight < 100 kg.
* Height 150-190 cm.
* Hip width between 30 - 45 cm.
* Distance from hip joint centre to knee joint centre: 36 cm - 50 cm.
* Distance from the centre of the knee joint to the ground: 43.5 - 59.5 cm.
* Shoe size EU 36-45.
* Patients must be able to follow simple commands.
* Age 18-85 years.
* Diagnosis of ABI or SCI.
* FAC level in participants with ABI < 4.
* WISCI II level in participants with SCI < 20.

Exclusion Criteria:

* Spasticity (MAS) = 4 in lower limbs.
* Skin alterations in the areas of contact with the device.
* Planned surgical intervention during the duration of the study.
* Two or more osteoporotic fractures in the lower limbs in the last 2 years.
* Presence of other pathologies causing exercise intolerance (such as uncontrolled hypertension, coronary artery disease, arrhythmia, congestive heart failure, severe pulmonary disease).
* Surgical operation in the 3 months prior to the start of the study on the limbs and/or spine.
* Psychiatric disorders that interfere with proper use of the device or participation in the study such as impulsivity or inability to understand simple commands.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | Through study completion, an average of 100 days
  Assessment of heart rate (beats/min)
Oxygen saturation | Through study completion, an average of 100 days
  % O2
Systolic blood pressure | Through study completion, an average of 100 days
  Assesment of systolic blood pressure in mmHg
Diastolic blood pressure | Through study completion, an average of 100 days
  Assesment of diastolic blood pressure in mmHg
Skin integrity | Through study completion, an average of 100 days
  Assess the size (centimetres) of the skin tag produced after use of the exoskeleton.
Pain (Visual Analogic Scale) | Through study completion, an average of 100 days
  Pain registered before and after the use of the device, by the participant and therapist. The options are from 1 to 6. A higher score means a worse outcome. Pain registered before and after the use of the device, by the participant and therapist. The options are from 1 to 6. A higher score means a worse outcome.
Fall prevalence | During the use of the device, for 6 weeks.
  Number of falling events ocurred from the participant or therapist.
Kinematic gait analysis | Once during the first session.
  Assessed by photogrammetry (VICON) in a gait analysis laboratory in healthy subjects
Muscular activation | Once during the first session.
  Assessed by electromyography (NORAXON).
Functional Ambulation Categories | In all sessions during 6 weeks.
  ABI participants
Walking Index for Spinal Cord Injury (WISCI) | In all sessions during 6 weeks.
  SCI participants
Time and assistance with device attachment and removal | In all sessions during 6 weeks.
  Time taken in minutes to fit and remove the participant's device.
Timed Up and Go (TUG) | In all sessions during 6 weeks.
  Distance to go 3 metres, turn around and sit on a chair.
6 Minutes Walking Test (6MWT) | In all sessions during 6 weeks.
  Distance covered using the device in 6 minutes
10 Meters Walking Test (10MWT) | In all sessions during 6 weeks.
  Time to cover 10 meters using the decvice.
Device malfunction | In all sessions during 6 weeks.
  Number and type of device malfunction
User perception of the device (QUEST 2.0) | At the end of the study, 6th week
  QUEST 2.0 will be assessed by the participant
Participant's satisfaction of the device (Participant Satisfaction scale). | At the end of the study, 6th week
  It will be measured through Participant Satisfaction scale.
Physiotherapist's satisfaction (Therapist Satisfaction Scale) | At the end of the study, 6th week
  It will be assessed using Therapist Satisfaction Scale
SF-12 | At the end of the study, 6th week
  Quality of life

SECONDARY OUTCOMES:
Acceptability | At the end of the study, 6th week
  Analysis of the drop-out rate during the study period.
Accesssibility | At the end of the study, 6th week
  Number of registered participants in relation to the data of potential participants who were not recruited obtained in the first screening

CONTACTS AND LOCATIONS:
Overall Officials: Elena García Armada, Dr., Principal Investigator — National Research Council
Locations (3):
- Spain (3):
  - CEADAC, Madrid
  - Centre for Automation and Robotics, Madrid
  - LESCER, Madrid

IPD SHARING:
Plan to Share IPD: No